CLINICAL TRIAL: NCT02300311
Title: A Multinational, Randomised, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Efficacy and Safety of Multiple Doses of Finalgon® Cream (1.08% Nicoboxil/ 0.17% Nonivamide) in the Treatment of Acute Low Back Pain
Brief Title: Efficacy and Safety of Finalgon® Cream Multiple Doses in Acute Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 69.53
Record Dates: First submitted 2014-11-24; First posted 2014-11-25 (Estimated); Results first posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-07

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — nonivamide; nicoboxil

ARMS (2):
- nonivamide + nicoboxil (Finalgon cream) (Experimental): 2 cm cream line for a skin area of approximately 20 x 20 cm2 up to 3 times in a 24h period
  Interventions: Drug: nonivamide + nicoboxil (Finalgon cream)
- placebo (Placebo Comparator): 2 cm cream line for a skin area of approximately 20 x 20 cm2 up to 3 times in a 24h period
  Interventions: Drug: placebo matching nonivamide + nicoboxil (Finalgon cream)

INTERVENTIONS:
Drug: nonivamide + nicoboxil (Finalgon cream) — 2 cm cream line for a skin area approximately 20 x 20 cm2 up to 3 times in a 24 hour period
  Arms: nonivamide + nicoboxil (Finalgon cream)
Drug: placebo matching nonivamide + nicoboxil (Finalgon cream) — 2 cm cream line for a skin area of approximately 20 x 20 cm2 up to 3 times in a 24h period
  Arms: placebo

SUMMARY:
To evaluate efficacy of Finalgon® cream (1.08% Nicoboxil/ 0.17% Nonivamide) versus placebo in patients with acute low back pain. To investigate the safety and tolerability of repeated use of Finalgon® cream (1.08% Nicoboxil/ 0.17% Nonivamide).

ELIGIBILITY:
Inclusion criteria:

1. Patients must sign and date an Informed Consent consistent with International Conference on Harmonisation (ICH)/Good Clinical Practice (GCP) guidelines and local regulation prior to participation in the trial.
2. Patients must agree to cooperate with all trial evaluations and perform all required tasks.
3. Patients must have acute nonspecific low back pain, ICD-10 code: M54.5.
4. Patients must have acute low back pain for more than 2 days and less than 21 days (= 3 weeks).
5. Male or female more or equal 18 and less or equal 65 years of age at Visit 1(Baseline).
6. Low back pain Pain intensity more or equal 5 on a 0-10 numerical rating scale (NRS).

Exclusion criteria:

1. Patients with a significant disease other than acute nonspecific low back pain. A significant disease is defined as a disease which, in the opinion of the investigator, may (i) put the patient at risk because of participation in the trial, or (ii) influence the results of the trial, or (iii) cause concern regarding the patient's ability to participate in the trial.
2. Multilocular pain or panalgesia.
3. History of more than 3 low back pain episodes in the last 6 months.
4. Acute low back pain due to vertebral collapse or neoplastic, inflammatory (ankylosing spondylitis), traumatic, or infective origins.
5. Abnormal findings in at least one of the following assessments: Achilles tendon reflex, patella reflex, heel walking, toe walking, cutaneous sensitivity of the legs (including gluteal region), paresis tests in supine position upon dorsiflexion, plantarflexion, hip flexion, knee extension.
6. Neurogenic Bladder and/or rectum dysfunction.
7. Any condition, disease or concomitant treatment that in the judgement of the investigator will affect the patient's ability to participate in the clinical trial or which will influence the trial methodology used.
8. Negative experience in the past with heat treatment for muscle complaints (e. g. hot water bottle, heat pads, hyperemisation-inducing topical creams, ointments or patches).
9. Patients with history of treatment of back pain with centrally acting drugs (e.g. opioids) and muscle relaxants within 6 months prior to enrolment.
10. Surgery due to back pain or rehabilitation due to back pain in the last 12 months.
11. Spinal injection back pain treatment within 6 months prior to enrolment.
12. Intake of antidepressant/antipsychotic medication within 4 weeks prior to enrolment.
13. Treatment of the recent low back pain period with oral analgesics for more than 4 consecutive days.
14. Locally applied medication to the back within 24 hours prior to enrolment (topical treatments, injections).
15. Non-pharmacological low back pain treatment (physiotherapy, heat treatment [e.g. hot water bottle, heat patch], or massages) within 12 hours prior to enrolment.
16. Administration of other analgesics within 12 h prior to enrolment (exception: acetylsalicylic acid [ASS] up to 100 mg/daily for anti-platelet-aggregation therapy).
17. Non-pharmacological low back pain treatment (physiotherapy, heat treatment [e.g. hot water bottle, heat patch], or massages) within 12 hours prior to enrolment.
18. Participation in an investigational drug or device trial within 4 weeks prior to enrolment.
19. History of treatment of back pain with centrally acting drugs (e.g. opioids) and muscle relaxants.
20. Treatment of the recent low back pain period with oral analgesics for more than 4 consecutive days.
21. Surgery due to back pain or rehabilitation due to back pain in the last 12 months.
22. Spinal injection back pain treatment within 6 months prior to enrolment.
23. Intake of antidepressant/antipsychotic medication within 4 weeks prior to enrolment.
24. Known hypersensitivity to nicoboxil, nonivamide, or other ingredients of the cream.
25. Known hypersensitivity to paracetamol.
26. Skin lesions (e.g. rash, bruising, laceration) in the back region.
27. Known history of central nervous system diseases with severe intellectual and memory disorders, psychiatric disorders.
28. History of abuse of alcohol/drugs within six months prior to enrolment.
29. Acute and relapsed chronic kidney diseases.
30. Severe hepatocellular insufficiency.
31. Pregnant or nursing women, including female patients with positive ß-HCG test at Visit 1.
32. Female patients of child-bearing potential not using highly effective method of birth control.
33. Patients who are currently participating in another trial or who have been participating in another trial within one month prior to Visit 1, and patients who have previously been randomised in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (8):
- Russia (6):
  - 69.53.53201 Boehringer Ingelheim Investigational Site, Kyiv
  - 69.53.53102 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 69.53.53103 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 69.53.53105 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 69.53.53106 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 69.53.53107 Boehringer Ingelheim Investigational Site, Saint Petersburg
- Ukraine (2):
  - 69.53.53202 Boehringer Ingelheim Investigational Site, Kyiv
  - 69.53.53203 Boehringer Ingelheim Investigational Site, Kyiv

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Multinational, multi-centre, randomised, double-blind, placebo-controlled, parallel group, 2-arm study with a treatment duration of up to 4 days
Groups:
- Placebo: Topical administration of Placebo cream. One application consists of 2 cm cream line for a skin area of approximately 20 x 20 square cm (corresponding to approximately 2 x hand size) up to 3 times in a 24 h period. Treatment duration consists of up to 4 days.
- Finalgon® Cream (Nicoboxil/ Nonivamide): Topical administration of Finalgon® cream (1.08% Nicoboxil/ 0.17% Nonivamide). One application consists of 2 cm cream line (3.5 mg Nicoboxil/ 0.5 mg Nonivamide) for a skin area of approximately 20 x 20 square cm (corresponding to approximately 2 x hand size) up to 3 times in a 24 h period.
  Treatment duration consists of up to 4 days.
Period: Overall Study
Arm/Group | Placebo | Finalgon® Cream (Nicoboxil/ Nonivamide)
Started | 69 | 69
Completed | 50 | 69
Not Completed | 19 | 0
Not completed — Other than the reason specified | 1 | 0
Not completed — Refused to continue taking medication | 18 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): All randomised patients who used at least one dose of study medication were included in the treated set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Finalgon® Cream (Nicoboxil/ Nonivamide) | Total
Number analyzed (Participants) | 69 | 69 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.52 (11.34) | 44.25 (12.68) | 43.38 (12.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 49 | 86
  Male | 32 | 20 | 52

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Difference (PID) From Pre-dose Baseline to 8h After the First Trial Medication Application (PID8h)
Description: Pain intensity (PI) was assessed on a 11-point numerical rating scale ranging from 0 (no pain) to 10 (worst pain possible) at pre-dose baseline and 0.5, 1, 2, 3, 4, 6 and 8 hours after trial medication application.
  The left side of each scale (0) is marked 'no pain' and the right side of the scale (10) is marked 'worst pain possible'.
  PID8h= Pain intensity (PI)8h - PI(baseline).
  Means reported are the adjusted means.
Time Frame: Baseline and 8 hours after trial medication application
Population: Full analysis set (FAS): All patients included in the treated set who provide any post-treatment data for the primary efficacy endpoint constituted the full analysis set.
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | Finalgon® Cream (Nicoboxil/ Nonivamide)
Number analyzed (Participants) | 69 | 69
points on a scale | -0.98 (0.215) | -2.82 (0.221)
Statistical Analysis 1: Comparison: Placebo vs Finalgon® Cream (Nicoboxil/ Nonivamide); PID8 utilised a restricted maximum likelihood (REML) based repeated measures approach, using all available longitudinal pain intensity observations at each post-baseline time up to 8 hours. The statistical model was applied to the analysis of change from baseline in pain intensity at 0.5, 1, 2, 3, 4, 6 and 8 hours; Test type: Superiority or Other; p < 0.0001, REML based repeated measures approach — The model included the fixed, categorical effects of treatment, country, time and treatment-by-time interaction and the continuous covariate of baseline PI; restricted maximum likelihood (REML) based repeated measures approach; Mean Difference (Final Values) = -1.849, 95% CI 2-sided [-2.454 to -1.244], Standard Error of Mean 0.306 — Differences between the treatment group effects (Finalgon® cream - placebo)

2. Secondary Outcome: Pain Intensity Difference (PID) From Pre-dose Baseline to 4 Hours After the First Trial Medication Application (PID4h)
Description: Pain intensity was assessed on a 11-point numerical rating scale ranging from 0 (no pain) to 10 (worst pain possible) at pre-dose baseline and 0.5, 1, 2, 3 and 4 hours after trial medication application. The left side of each scale (0) is marked 'no pain' and the right side of the scale (10) is marked 'worst pain possible'. PID4h= PI(4h) - PI(baseline). Means reported are the adjusted means.
Time Frame: Baseline and 4 hours after trial medication application
Population: as for outcome 1
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | Finalgon® Cream (Nicoboxil/ Nonivamide)
Number analyzed (Participants) | 69 | 69
points on a scale | -0.77 (0.157) | -2.11 (0.196)
Statistical Analysis 1: Comparison: Placebo vs Finalgon® Cream (Nicoboxil/ Nonivamide); PID4 utilised a restricted maximum likelihood (REML) based repeated measures approach, using all available longitudinal pain intensity observations at each post-baseline time up to 4 hours. The statistical model was applied to the analysis of change from baseline in pain intensity at 0.5, 1, 2, 3, and 4 hours; Test type: Superiority or Other; p < 0.0001, REML based repeated measures approach — The statistical model included the fixed, categorical effects of treatment, country, time and treatment-by-time interaction and the continuous covariate of baseline PI; restricted maximum likelihood (REML) based repeated measures approach; Mean Difference (Final Values) = -1.341, 95% CI 2-sided [-1.832 to -0.851], Standard Error of Mean 0.248 — Differences between the treatment group effects (Finalgon® cream - placebo)

3. Secondary Outcome: Difference of Average Pain Intensity (APID) From Pre-dose Baseline on the Last Individual Treatment Day
Description: Difference of average pain intensity from pre-dose baseline on the last individual treatment day (The last individual treatment day was the last day on which the patient had recorded the study drug applications within the patient diary). Pain intensity was assessed by the patient using 0-10 numerical rating scale (NRS).
  Patients were given two 0-10 numerical rating scales (NRS) - to self-report of pain intensity at given time points for the period 0-8 hours post first dose and to self-report of average pain intensity they had at each treatment day. The left side of each scale (0) is marked 'no pain' and the right side of the scale (10) is marked 'worst pain possible'. APIDtime point = APItime point - PI baseline (time point is the last individual treatment day (either Day 1, 2, 3 or 4 after drug administration)).
  Means reported are the adjusted means.
Time Frame: Baseline and 1 to 4 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | Finalgon® Cream (Nicoboxil/ Nonivamide)
Number analyzed (Participants) | 69 | 69
points on a scale | -2.17 (0.272) | -5.13 (0.279)
Statistical Analysis 1: Comparison: Placebo vs Finalgon® Cream (Nicoboxil/ Nonivamide); The difference of average pain intensity from pre-dose baseline on the last individual treatment day was analysed using ANCOVA; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA using the fixed, categorical effects of treatment and country as well as the continuous covariate of baseline PI; Mean Difference (Final Values) = -2.958, 95% CI 2-sided [-3.712 to -2.205], Standard Error of Mean 0.381 — Differences between the treatment group effects (Finalgon® cream - placebo)

4. Secondary Outcome: Patient's Assessment of the Efficacy on the Last Individual Treatment Day
Description: Patients were asked to rate the effect of the study medication for relieving their low back pain using a 4-point verbal rating scale (1=Poor, 2= Fair, 3=Good, 4=Very Good).
Time Frame: 1 to 4 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Finalgon® Cream (Nicoboxil/ Nonivamide)
Number analyzed (Participants) | 69 | 69
percentage of participants
  Very good | 13.0 (0.272) | 29.0 (0.279)
  Good | 17.4 | 58.0
  Fair | 20.3 | 13.0
  Poor | 47.8 | 0.0
  Missing | 1.4 | 0.0
Statistical Analysis 1: Comparison: Placebo vs Finalgon® Cream (Nicoboxil/ Nonivamide); For the analysis of the repeated multinomial efficacy endpoint 'patient assessment of efficacy' on the last individual treatment day, ordinal logistic regression models is used. Only non-missing data is analysed in the statistical model; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Ordinal logistic regression models adjusting for the continuous covariate 'baseline PI' and the categorical variable 'country' was performed; Odds Ratio (OR) = 11.370, 95% CI 2-sided [5.342 to 24.199] — Odds ratio of (Finalgon® cream / placebo)

ADVERSE EVENTS:
Time Frame: Adverse Event's collected after the first dose and upto the residual effect period (REP) period after the last drug administration (from first study administration until 24 hours after last study administration) ie. up to 5 days.
Arm/Group | Placebo | Finalgon® Cream (Nicoboxil/ Nonivamide)
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/69
Other Adverse Events (participants affected / at risk) | 0/69 | 0/69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights